CLINICAL TRIAL: NCT04063384
Title: Subjective Response to Alcohol and Associated Neural Systems in Bipolar Disorder
Brief Title: Acute Alcohol Response In Bipolar Disorder: a fMRI Study
Acronym: BACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Elizabeth Thomas Cox Lippard, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: K01AA027573 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-21 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder; Alcohol Drinking; Alcohol Use Disorder
MeSH Terms: conditions — Bipolar Disorder; Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Active Comparator): Participants will be dosed to a 0.08g% blood alcohol concentration.
  Interventions: Other: alcohol beverage
- Placebo (Placebo Comparator): Participants will receive a low dose of alcohol (placebo condition).
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Other: alcohol beverage — Participants will be provided alcohol during study visits and changes in behavior/neural activity after consuming alcohol will be examined.
  Arms: Alcohol
Other: Placebo beverage — placebo beverage conditions.
  Arms: Placebo

SUMMARY:
Alcohol use disorders (AUDs) affect up to 60% of individuals with bipolar disorder during their lifetime-a rate 3 to 5 times higher than what occurs in the general population. The mechanisms that contribute to elevated rates of comorbidity are not known. Early identification in individuals with bipolar disorder who are at risk for AUDs could inform novel intervention strategies and improve life-long outcomes. The primary objective of this protocol is to use alcohol administration procedures and functional MRI techniques to investigate subjective response to alcohol, compared to placebo, and relationship with functional responses of, and connectivity among, brain regions in ventral prefrontal emotional networks in young adults with bipolar disorder and healthy comparison young adults. Baseline clinical and structural MRI assessments will be completed in 30 bipolar and 30 healthy young adults (21-26 years of age, 50% women). Then, following standard beverage administration procedures, participants will complete within-person, counter-balanced, fMRI scans and complete measures of subjective response to alcohol while under the influence of alcohol or placebo. Specifically, individual differences in the experience of stimulating, sedative, and anxiolytic effects of alcohol (measured with self-report surveys) and individual differences in neural responses to alcohol within ventral prefrontal emotional networks will be investigated and differences in bipolar disorder compared to healthy participants assessed. Functional MRI scans during a continuous performance task with emotional and neutral distractors (CPT-END) and at rest will be collected while under the influence of alcohol and placebo and compared. Experience of stimulating, sedative, and anxiolytic effects of alcohol from self-report survey data and neural responses to emotional stimuli while under the influence of alcohol compared to placebo will be the primary data outcomes assessed. Additionally, associations between subjective and neural response to alcohol and drinking patterns will be explored (secondary outcomes). The primary endpoint of the study will be after completion of both alcohol and placebo beverage conditions.

DETAILED DESCRIPTION:
A total of 60 bipolar and healthy comparison subjects (n=30 per group, 21-26 years of age, 50% women, with no history of a moderate/severe AUD) will be recruited from the greater Austin area. Once recruited and enrolled, subjects will undergo detailed structured clinical evaluations to verify inclusion and exclusion criteria, comprehensive assessment of alcohol and other drug use history, and cognitive testing, followed by structural MRI assessments. Following standard beverage administration procedures, they will then complete measures of subjective response to alcohol and fMRI scans while under the influence of alcohol or a placebo condition (counter-balanced). For each participant the first beverage session assignment (whether the participant is given alcohol or the placebo beverage first) will be randomized. Alcohol and placebo sessions will occur within 3 days of each other. FMRI assessments will include a continuous performance task with emotional and neutral distractors (CPT-END) and a resting state scan.

For both the alcohol and the placebo beverage conditions, the protocol will be the same. The beverage administration sessions will occur in a private room at the University of Texas at Austin in the Imaging Research Center. The table in the testing room will be wiped down with alcohol prior to the participant's arrival (olfactory cue). Study staff will use an algorithm to calculate individual alcohol doses based on the participants' age, sex, height, and weight. Participants fast from food for 4 hours prior to their session. Before beginning consumption of their beverages, they will eat a weight-adjusted, 1 calorie per pound snack of pretzels. While participants eat their pretzels, study staff will mix beverages in front of participants. Vodka and placebo (decarbonated tonic water) will be stored in absolute vodka bottles, measured out, and combined with mixer in front of participants. Mixed drinks will be poured into glasses that have been sitting face down with rims soaking in vodka. Prior to giving the beverage to the participant, all drinks will get an alcohol floater (squirt of absolute vodka on top of the drink). Participants will be given 20 minutes to orally consume two beverages (10 minutes per beverage).

Following oral consumption and a 10 minute absorption period, breathalyzer tests will be conducted to identify a .06g% ascending limb breath alcohol concentration (BrAC). Self-report of subjective response to alcohol will be collected and participants will immediately enter the scanner and complete the fMRI scan (acquisition parameters are identical during alcohol and placebo conditions). BrAC will be tracked after the MRI scan and subjective response to alcohol collected again at peak BrAC and at descending BrAC of .06g%. Consistent with NIAAA guidelines for human alcohol studies, BrAC readings will continue every 30 minutes until participants are below 0.04% at which time they will be escorted home. During the placebo condition, participants will be given false BrAC readings. False BrAC readings given to participants during the placebo session will be based on the average BrACs we record during the alcohol sessions. The average time participants stay in the laboratory will be the same for the placebo and alcohol beverage conditions. Participants are debriefed after completing all sessions and the need for deception to ensure the placebo-controlled alcohol session will be explained.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants:

* between 21 and 26 years of age
* having consumed at least 4 (men) or 3 (women) drinks on a single occasion over the last year
* euthymic at the time of study

Inclusion criteria for bipolar disorder participants:

- Meeting Diagnostic and Statistical Manual-5 Research Version (DSM-V-RV) diagnostic criteria for bipolar disorder, confirmed by structured interview

Exclusion Criteria:

For all subjects exclusion criteria include:

* history of significant medical illness, particularly if possible changes in cerebral tissue
* neurologic abnormality including significant head trauma (loss of consciousness of ≥5-min)
* full Scale intelligence quotient (IQ) <85
* contraindication to MRI scanning
* positive pregnancy test
* current cannabis use disorder>moderate
* history of severe AUDs
* scores > 15 on the alcohol Use Disorders Identification Test (AUDIT; part of phone screen)
* ever being in an abstinence-oriented treatment program for alcohol use
* reporting wanting to quit drinking but not being able to
* any medical, religious, or other reasons for not drinking alcohol
* history of heart attack, heart trouble, high blood pressure, diabetes, or liver disease
* an adverse reaction to alcoholic beverages
* reporting never consuming 4 (men) or 3 (women) or more drinks on a single occasion over the last year
* unwillingness to have a friend or family member drive them home after the alcohol administration sessions
* a past year substance use disorder (other than alcohol, cannabis, or nicotine)

Additional exclusion criteria for bipolar disorder participants:

- not taking medications for greater than or equal to 4 weeks (i.e. participants must be stable on medications)

Additional exclusion criteria for healthy comparison subjects also include:

* any prior psychiatric hospitalizations
* lifetime history of a neurodevelopmental disorder, affective disorder, psychotic disorder, eating disorder
* greater than 1 month of lifetime psychotropic medication. -

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lippard, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion and publication of finding, functional neuroimaging data and behavior data collected following alcohol and placebo conditions will be shared.
Supporting Information: SAP
Time Frame: We will complete all our analyses and publish results and methodologies in scientific journals before the data are available to the research community. Data will be made available following 6 months after publication.
Access Criteria: We will be collecting identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Result] Kirsch DE, Kosted R, Le V, Almeida JRC, Fromme K, Strakowski SM, Lippard ETC. Ventral prefrontal network response to alcohol in young adults with bipolar disorder: a within-subject randomized placebo-controlled alcohol administration study. Neuropsychopharmacology. 2023 Dec;48(13):1910-1919. doi: 10.1038/s41386-023-01657-6. Epub 2023 Jul 20. PMID 37474761
- [Result] Kosted R, Kirsch DE, Le V, Fromme K, Lippard ETC. Subjective response to alcohol: Interactive effects of early life stress, parental risk for mood and substance use disorders, and drinking context. Pharmacol Biochem Behav. 2023 Aug;229:173591. doi: 10.1016/j.pbb.2023.173591. Epub 2023 Jun 22. PMID 37353164
- [Result] Lippard ETC, Kirsch DE, Kosted R, Le V, Almeida JRC, Fromme K, Strakowski SM. Subjective response to alcohol in young adults with bipolar disorder and recent alcohol use: a within-subject randomized placebo-controlled alcohol administration study. Psychopharmacology (Berl). 2023 Apr;240(4):739-753. doi: 10.1007/s00213-023-06315-9. Epub 2023 Jan 25. PMID 36695842
- [Result] Kirsch DE, Le V, Kosted R, Fromme K, Lippard ETC. Neural underpinnings of expecting alcohol: Placebo alcohol administration alters nucleus accumbens resting state functional connectivity. Behav Brain Res. 2023 Feb 2;437:114148. doi: 10.1016/j.bbr.2022.114148. Epub 2022 Oct 4. PMID 36206822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 participants were recruited.
Pre-assignment Details: Participants were randomly assigned to receiving placebo first or alcohol beverage session first.
Groups:
- BD Alcohol First, Then Placebo; TD Alcohol First, Then Placebo: Participants will be dosed to a 0.08g% blood alcohol concentration on alcohol day and then on a following day was dosed to <.01 blood alcohol concentration (placebo day).
- BD Placebo First, Then Alcohol; TD Placebo First, Then Alcohol: Participants were dosed to <.01 blood alcohol concentration (placebo day) for their first beverage, and then on a following day were dosed to a 0.08g% blood alcohol concentration (alcohol day).
Period: Overall Study
Arm/Group | BD Alcohol First, Then Placebo | TD Alcohol First, Then Placebo | BD Placebo First, Then Alcohol | TD Placebo First, Then Alcohol
Started | 16 | 15 | 14 | 15
Completed | 15 | 13 | 13 | 14
Not Completed | 1 | 2 | 1 | 1
Not completed — placebo manipulation issue | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants with placebo manipulation issues were excluded from analysis. One participant in the TD group later revealed a past depressive episode and was excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | BD Alcohol First, Then Placebo | TD Alcohol First, Then Placebo | BD Placebo First, Then Alcohol | TD Placebo First, Then Alcohol | Total
Number analyzed (Participants) | 15 | 13 | 13 | 13 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (1.8) | 22.1 (1.3) | 23.5 (1.7) | 22.9 (1.3) | 22.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 7 | 35
  Male | 4 | 5 | 4 | 6 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4 | 3 | 7 | 3 | 17
  Nonhispanic White | 10 | 6 | 3 | 4 | 23
  Asian | 0 | 3 | 2 | 5 | 10
  More than one race | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Level of Intoxication (Subjective Response) on Each Condition Day After Drinking Relative to How They Felt When Arriving to the Lab on That Respective Day )Prior to Drinking)
Description: Participants fill out self-report surveys [specifically the Subjective Effects of Alcohol Scale (SEAS)] on how they feel when they arrive to their beverage administration sessions (alcohol and placebo sessions). They then feel out the same self-report surveys on how intoxicated they feel during their beverage sessions (alcohol and placebo). Changes in how intoxicated they feel is calculated for both the alcohol and placebo condition (compared to how they felt pre-beverage). 4 subscores are calculated by summing individual items: positive valence/positive arousal (stimulation), SEAS positive valence/negative arousal (anxiolytic), negative valence/negative arousal (aggression/agitation), and negative valence/negative arousal (sedative effects). Summed subscores on the SEAS range between 0 and 40. Change scores can therefore range between -40 and 40 (post-beverage compared to pre-beverage feelings). Scores greater than 0 on any one subscale indicates feeling more effects of alcohol.
Time Frame: up to 1 week
Population: Excluded participants with placebo manipulation issues. One TD participant was excluded because they later revealed a past depressive episode.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BD Alcohol First, Then Placebo | TD Alcohol First, Then Placebo | BD Placebo First, Then Alcohol | TD Placebo First, Then Alcohol
Number analyzed (Participants) | 15 | 13 | 13 | 13
score on a scale
  SEAS positive valence/positive arousal: alcohol session | 7.3 (1.2) | 3.6 (1.0) | 15.4 (2.3) | 6.3 (1.3)
  SEAS positive valence/positive arousal: placebo session | 4.1 (1.1) | 2.3 (0.98) | 5.3 (1.8) | 3.3 (1.1)
  SEAS positive valence/negative arousal: alcohol session | -1.4 (1.6) | -5.3 (0.9) | 7.1 (2.1) | 0.9 (1.4)
  SEAS positive valence/negative arousal: placebo session | 1.7 (0.98) | -0.42 (0.47) | -2.3 (0.97) | -2.96 (4.7)
Statistical Analysis 1: Comparison: BD Alcohol First, Then Placebo vs TD Alcohol First, Then Placebo vs BD Placebo First, Then Alcohol vs TD Placebo First, Then Alcohol; Test type: Other; p < 0.05, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons; Group (bipolar, healthy)-by-condition (alcohol, placebo)-by-time of subjective response interactions on subjective response to alcohol were modeled, covarying beverage condition order, biological sex, and age, with SEAS and DEQ subscale scores as the dependent variables. Time of subjective response (pre- and post-scan) and beverage condition (alcohol, placebo) were within-subject factors and group was an independent between-subject factor

2. Primary Outcome: Change in Functional Coupling Between Regions of Interest During Viewing of Emotional Stimuli (Neural Responses While Viewing Emotional Stimuli Were Contrasted Against Neural Responses When Viewing Squares)
Description: Neural responses to emotional stimuli during the alcohol and placebo sessions were modeled. Fisher transformed correlation coefficients between regions of interest while viewing emotional stimuli (compared to squares) were calculated for each beverage session and data extracted for posthoc analysis. Values represent change scores in correlation coefficients during each beverage session.
Time Frame: up to 1 week
Population: Analysis was completed prior to study completion.
Measure: Mean (Standard Error); unit: Change scores in correlation coefficient
Arm/Group | BD Alcohol First, Then Placebo | TD Alcohol First, Then Placebo | BD Placebo First, Then Alcohol | TD Placebo First, Then Alcohol
Number analyzed (Participants) | 11 | 12 | 12 | 13
Change scores in correlation coefficient
  Insula:sgACC functional connectivity: alcohol | -0.04 (0.02) | 0.03 (0.02) | 0.002 (0.02) | 0.05 (0.03)
  Insula:sgACC functional connectivity: placebo | 0.001 (0.02) | -0.0003 (0.02) | 0.05 (0.01) | -0.006 (0.02)
  Left NAc:vmPFC functional connectivity: alcohol | -0.006 (0.03) | -0.05 (0.02) | 0.01 (0.02) | -0.02 (0.03)
  Left NAc:vmPFC functional connectivity: placebo | -0.06 (0.02) | -0.002 (0.02) | -0.014 (0.03) | 0.003 (0.02)
Statistical Analysis 1: Comparison: BD Alcohol First, Then Placebo vs TD Alcohol First, Then Placebo vs BD Placebo First, Then Alcohol vs TD Placebo First, Then Alcohol; Power analysis suggests this sample size (n = 23 with bipolar disorder, n = 24 healthy comparison participants), at an alpha = 0.05, provides > 80% statistical power to detect a within subject effect size (ES) d ≥ 0.6 in both subgroups and a between group ES d ≥ 0.8 in this fMRI analysis; Test type: Other; p < 0.004, Mixed Models Analysis — Results of primary models were considered significant at p ≤ 0.004 (Bonferroni correction for twelve ROI-to-ROI connections); We used a mixed model to examine group by condition by hemisphere (left, right) interactions on ROI-to-ROI FC response to emotional stimuli (contrast: emotional stimuli - squares). Group was an independent between-subject factor, condition and hemisphere were within-subject factors, and ROI-to-ROI FC was the dependent variable

ADVERSE EVENTS:
Time Frame: Adverse event data was collected following enrollment and through completion of both beverage sessions.
Description: This did not differ from the clinicaltrials.gov definitions.
Groups:
- BD Alcohol First; TD Alcohol First: Participants will be dosed to a 0.08g% blood alcohol concentration on their first beverage day
- BD Placebo First; TD Placebo First: Participants were dosed to <.01 blood alcohol concentration (placebo day) for their first beverage
- BD Alcohol Second; TD Alcohol Second: Participants will be dosed to a 0.08g% blood alcohol concentration on their second beverage day
- BD Placebo Second; TD Placebo Second: Participants were dosed to <.01 blood alcohol concentration (placebo day) for their second beverage
Arm/Group | BD Alcohol First | TD Alcohol First | BD Placebo First | TD Placebo First | BD Alcohol Second | TD Alcohol Second | BD Placebo Second | TD Placebo Second
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Drinking was performed in a clinical space and lacks ecological validity (representing real world drinking environment). How individuals reported feeling may not generalize to how they feel when they consume alcohol regularly. Additionally, participants were the only one drinking. Individuals may respond differently when drinking in more social environments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT04063384/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04063384/ICF_002.pdf